CLINICAL TRIAL: NCT00810277
Title: An Open Label Study to Evaluate the Safety and Effect on Disease Activity of Tocilizumab in Patients With Active Rheumatoid Arthritis on Background Non-biologic DMARDs Who Have an Inadequate Response to Current Non-biologic DMARDs.
Brief Title: A Study of Tocilizumab in Patients With Rheumatoid Arthritis Who Have an Inadequate Response to Current Non-Biologic DMARDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22012; 2008-004126-16
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks for 24 weeks

SUMMARY:
This single arm study will assess the safety and efficacy of tocilizumab in patients with moderate to severe active rheumatoid arthritis who have an inadequate response to current non-biologic DMARDs. Patients will receive iv infusions of tocilizumab 8mg/kg every 4 weeks for a total of 6 infusions, either as monotherapy or in combination with their current non-biologic DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* moderate to severe rheumatoid arthritis;
* inadequate response to current non-biologic DMARDs

Exclusion Criteria:

* rheumatic autoimmune disease or inflammatory joint disease other than rheumatoid arthritis;
* previous treatment with other biologics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11-30 (Actual); Primary Completion 2010-05-26 (Actual); Study Completion 2010-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Finland (3):
  - Kanta-Hämeen Keskussairaala ; Reumatologia, Hämeenlinna
  - Kiljavan Lääketutkimus Oy, Hyvinkää
  - Kanta-Hämeen keskussairaala; Riihimäen aluesairaala Reumapoliklinikka, Riihimäki

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab at a dose of 8 milligram per kilogram (mg/kg) via intravenous infusion every 4 weeks up to 24 weeks.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 14
Completed | 13
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who entered the study.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.86 (9.662)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both serious as well as non-serious AEs.
Time Frame: Baseline up to Week 24
Population: Analysis population included all participants who entered the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
percentage of participants
  AEs | 92.9
  SAEs | 7.1

2. Secondary Outcome: Disease Activity Score (DAS28)
Description: DAS28 was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joints count, erythrocyte sedimentation rate (ESR) (mm/hour) or C-reactive protein (CRP) (mg/dL), and general health (GH) status (measured on a 0 to 100 mm Visual Analogue Scale [VAS] where 0=no disease activity and 100=worst disease activity). DAS28 was calculated using following formulas: DAS28-ESR = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*GH of disease activity; DAS28-CRP = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(10*CRP+1) + 0.014*GH of disease activity. DAS28-ESR was adopted to calculate DAS28 if effective ESR data was available; otherwise DAS28-CRP was adopted to calculate DAS28. Total score range: 0-10, higher score=more disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Analysis population included all participants who entered the study. 'n'=number of participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
units on a scale
  DAS28 ESR: Baseline (n=14) | 5.9896986 (1.0636917)
  DAS28 ESR: Week 4 (n=14) | 2.852859 (1.3154333)
  DAS28 ESR: Week 8 (n=13) | 2.1529895 (1.0578132)
  DAS28 ESR: Week 12 (n=12) | 1.9199257 (0.9622713)
  DAS28 ESR: Week 16 (n=13) | 1.6475303 (1.205548)
  DAS28 ESR: Week 20 (n=13) | 1.6527143 (0.9999803)
  DAS28 ESR: Week 24 (n=13) | 1.977934 (1.5634882)
  DAS28 CRP: Baseline (n=14) | 5.7627144 (0.9613441)
  DAS28 CRP: Week 4 (n=14) | 3.3564332 (1.2154714)
  DAS28 CRP: Week 8 (n=13) | 2.684394 (0.9556779)
  DAS28 CRP: Week 12 (n=12) | 2.5826295 (1.0084694)
  DAS28 CRP: Week 16 (n=13) | 2.3791197 (1.0837377)
  DAS28 CRP: Week 20 (n=13) | 2.2859272 (1.0212892)
  DAS28 CRP: Week 24 (n=13) | 2.3343281 (1.2686423)

3. Secondary Outcome: Percentage of Participants Achieving DAS28 Remission (DAS28 <2.6)
Description: DAS28 was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) or CRP (mg/dL), and general health (GH) status (measured on a 0 to 100 mm Visual Analogue Scale [VAS] where 0=no disease activity and 100=worst disease activity). DAS28 was calculated using following formulas: DAS28-ESR = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*GH of disease activity; DAS28-CRP = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(10*CRP+1) + 0.014*GH of disease activity. DAS28-ESR was adopted to calculate DAS28 if effective ESR data was available; otherwise DAS28-CRP was adopted to calculate DAS28. Total score range: 0-10, higher score=more disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
percentage of participants
  DAS28 ESR: Week 4 (n=14) | 42.86
  DAS28 ESR: Week 8 (n=13) | 69.23
  DAS28 ESR: Week 12 (n=12) | 83.33
  DAS28 ESR: Week 16 (n=13) | 76.92
  DAS28 ESR: Week 20 (n=13) | 84.62
  DAS28 ESR: Week 24 (n=13) | 69.23
  DAS28 CRP: Week 4 (n=14) | 35.71
  DAS28 CRP: Week 8 (n=13) | 46.15
  DAS28 CRP: Week 12 (n=12) | 41.67
  DAS28 CRP: Week 16 (n=13) | 61.54
  DAS28 CRP: Week 20 (n=13) | 76.92
  DAS28 CRP: Week 24 (n=13) | 61.54

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20% (ACR20), ACR50 and ACR70 Response
Description: ACR20, ACR50, and ACR70 response: greater than or equal to (>=) 20 percent (%), 50%, and 70% improvement respectively, in tender or swollen joint counts and in 3 of the following criteria: (1) Participant's assessment of pain (measured on a 0 to 100 mm VAS where 0=no pain and 100=unbearable pain); (2) Participant's assessment of disease activity (measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity); (3) Investigator's global assessment of disease activity (measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity); (4) Participant's assessment of functional disability via health assessment questionnaire (HAQ) (measured using 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
percentage of participants
  ACR20: Week 4 (n=14) | 57.14
  ACR20: Week 8 (n=13) | 100.00
  ACR20: Week 12 (n=13) | 76.92
  ACR20: Week 16 (n=13) | 100.00
  ACR20: Week 20 (n=13) | 84.62
  ACR20: Week 24 (n=13) | 100.00
  ACR50: Week 4 (n=14) | 28.57
  ACR50: Week 8 (n=13) | 76.92
  ACR50: Week 12 (n=13) | 61.54
  ACR50: Week 16 (n=13) | 76.92
  ACR50: Week 20 (n=13) | 76.92
  ACR50: Week 24 (n=13) | 61.54
  ACR70: Week 4 (n=14) | 0.00
  ACR70: Week 8 (n=13) | 46.15
  ACR70: Week 12 (n=13) | 30.77
  ACR70: Week 16 (n=13) | 46.15
  ACR70: Week 20 (n=13) | 53.85
  ACR70: Week 24 (n=13) | 61.54

5. Secondary Outcome: C-Reactive Protein (CRP) Level
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
milligram per liter (mg/L)
  Baseline (n=14) | 35.81 (19.459)
  Week 4 (n=14) | 1.29 (0.994)
  Week 8 (n=13) | 1.43 (0.910)
  Week 12 (n=12) | 1.16 (0.700)
  Week 16 (n=13) | 2.42 (3.486)
  Week 20 (n=13) | 1.10 (0.648)
  Week 24 (n=13) | 2.96 (3.577)

6. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: The erythrocyte sedimentation rate (ESR) is the rate at which red blood cells sediment in a period of one hour.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter per hour (mm/h)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
millimeter per hour (mm/h)
  Baseline (n=14) | 37.14 (18.102)
  Week 4 (n=14) | 3.71 (3.832)
  Week 8 (n=13) | 4.85 (8.543)
  Week 12 (n=12) | 2.42 (0.996)
  Week 16 (n=13) | 3.00 (2.677)
  Week 20 (n=13) | 2.46 (1.050)
  Week 24 (n=13) | 6.46 (7.666)

7. Secondary Outcome: Percentage of Participants Who Discontinued the Study
Time Frame: Up to Week 24
Population: Analysis population included all participants who entered the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
percentage of participants | 7.1

8. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) Level Elevation More Than 1.5 Times Upper Limit of Normal
Description: Normal range of ALT is 7 to 56 units per liter (U/L) of serum. Normal range of AST is 5 to 40 units per liter (U/L) of serum.
Time Frame: Up to Week 24
Population: Analysis population included all participants who entered the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
percentage of participants
  >1.5 ULN ALT | 7.14
  >1.5 ULN AST | 7.69

9. Secondary Outcome: Percentage of Participants With Lipid Level Elevations
Description: Low density lipoprotein (LDL) level was categorized as 'Optimal (less than [<] 100 milligram per deciliter [mg/dL])', 'Near Optimal/Above Optimal (100-129 mg/dL)', 'Borderline High (130-159 mg/dL)', 'High (160-189 mg/dL)', and 'Very high (190 mg/dL)'. High density lipoprotein (HDL) level was categorized as 'Acceptable (40-59 mg/dL)', 'High (>=60 mg/dL)'. Total cholesterol (TC) level was categorized as 'Desirable (<200 mg/dL)', 'Borderline High (200-239 mg/dL)', 'High (>=240 mg/dL)'.
Time Frame: Week 24
Population: Analysis population included all participants who entered the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
percentage of participants
  LDL: Optimal | 15.38
  LDL: Near Optimal/Above Optimal | 30.77
  LDL: Borderline High | 38.46
  LDL: High | 15.38
  LDL: Very high | 0.00
  HDL: Acceptable | 30.77
  HDL: High | 69.23
  TC: Desirable | 30.77
  TC: Borderline High | 30.77
  TC: High | 38.46

10. Secondary Outcome: Neutrophil Count
Time Frame: Baseline, Weeks 4, 8, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: E^9 per liter
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
E^9 per liter
  Baseline (n=13) | 5.53 (1.849)
  Week 4 (n=14) | 2.31 (0.971)
  Week 8 (n=13) | 2.32 (1.059)
  Week 12 (n=11) | 2.12 (0.675)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=14)
Erysipelas (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=14)
Neutropenia (Blood and lymphatic system disorders) | 3
Arrhythmia (Cardiac disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Influenza like illness (General disorders) | 1
Infusion related reaction (General disorders) | 3
Gastroenteritis (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 1
Oral infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Blood cholesterol increased (Investigations) | 2
Blood potassium decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Lipids increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 2
Transaminases increased (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.